CLINICAL TRIAL: NCT03277638
Title: Phase I/II Study of Laser Interstitial Thermotherapy (LITT) Combined With Checkpoint Inhibitor for Recurrent GBM (RGBM)
Brief Title: Laser Interstitial Thermotherapy (LITT) Combined With Checkpoint Inhibitor for Recurrent GBM (RGBM)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3316; NCI-2017-02417 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma, Adult
Keywords: recurrent glioblastoma; brain cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Lead; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Three parallel groups given Pembrolizumab injections at different timepoints
Masking Description: Because this is an open-label, safety and tolerability study in which all enrolled subjects will receive Pembrolizumab in Combination with LITT, this study is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pembrolizumab injections 7 days before surgery (Experimental): Patients will have intravenous pembrolizumab 7 days before surgery with Laser Interstitial Thermotherapy
  Interventions: Drug: Pembrolizumab at 7 days prior; Procedure: Laser Interstitial Thermotherapy
- Pembrolizumab injections 14 days after surgery (Experimental): Patients will have intravenous pembrolizumab 14 days after surgery with Laser Interstitial Thermotherapy
  Interventions: Drug: Pembrolizumab at 14 days post; Procedure: Laser Interstitial Thermotherapy
- Pembrolizumab injections 35 days after surgery (Experimental): Patients will have intravenous pembrolizumab 35 days after surgery with Laser Interstitial Thermotherapy
  Interventions: Drug: Pembrolizumab at 35 days post; Procedure: Laser Interstitial Thermotherapy

INTERVENTIONS:
Drug: Pembrolizumab at 7 days prior — Pembrolizumab injections 7 days before surgery
  Other Names: Pembrolizumab
  Arms: Pembrolizumab injections 7 days before surgery
Drug: Pembrolizumab at 14 days post — Pembrolizumab injections 14 days after surgery
  Other Names: Pembrolizumab
  Arms: Pembrolizumab injections 14 days after surgery
Drug: Pembrolizumab at 35 days post — Pembrolizumab injections 35 days after surgery
  Other Names: Pembrolizumab
  Arms: Pembrolizumab injections 35 days after surgery
Procedure: Laser Interstitial Thermotherapy — surgical procedure to heat hard to reach tumors with a laser beam
  Other Names: LITT

SUMMARY:
The purpose of this study is to test the side effects and efficacy of using Laser Interstitial Thermotherapy (LITT) combined with Pembrolizumab. LITT is a minimally invasive surgical technique that uses a laser to heat brain tumors.

Pembrolizumab is an investigational (experimental) drug that works by helping participants' immune system work correctly to detect and fight cancer cells. Pembrolizumab is experimental because it is not approved by the Food and Drug Administration (FDA), for this use, though it is approved to treat other cancers.

DETAILED DESCRIPTION:
Primary Objectives:

1. Phase I: To determine the optimal timing for combining LITT and pembrolizumab in patients with rGBM:

   • To determine the feasibility, safety, tolerability and side effect profiles for combining LITT and pembrolizumab at various time points pre-LITT vs. post-LITT (Phase I).
2. Phase II: To estimate the response to pembrolizumab combined with LITT in patients with rGBM;

   • To estimate the response rate after treatment with LITT combined with pembrolizumab in patients with rGBM (Phase II).
3. To collect and record the side effect profiles for combining LITT and pembrolizumab (Phase I and Phase II).

Secondary Objectives:

1. To determine the effect of pembrolizumab on systemic immune microenvironment in patients with rGBM.
2. To determine the effect of pembrolizumab on the intra-tumoral immunosuppressive microenvironment within rGBM.
3. Secondary for Phase II, to estimate progression free survival (PFS) and overall survival (OS) after treatment with LITT combined with pembrolizumab in patients with rGBM (Phase II).
4. Measure radiological response using both conventional RANO criterion, a modified RANO (RANOi) designed specifically for immunotherapy response assessment, as well as MRI fingerprinting (MRF), recently demonstrated by the PI and collaborators to accurately and precisely distinguish recurrent GBM from radiation injury.
5. Correlate clinical and radiological response to known biomarkers of GBM such as Isocitrate Dehydrogenase 1 (IDH-1) mutations, Isocitrate Dehydrogenase 2 (IDH-2) mutations, Methyl-Guanine Methyl Transferase (MGMT) promoter methylation, Phosphatase and tensin homologue (PTEN) loss and KI-67.

Study Design:

The Phase I component will involve up to two of a possible 3 cohorts of 3-4 patients each for a total of 6-8 evaluable patients. Each patient will undergo a stereotactic biopsy. If GBM or Gliosarcoma is confirmed by frozen section, patients will undergo LITT then treatment with 200 mg pembrolizumab IV. Cohort I will receive pembrolizumab on post operative day 14 and every 3 weeks thereafter. In the event that one patient suffers non-hematologic toxicity of grade 3 or more, or if hematologic toxicity is grade 4 or higher, the investigators will delay the 2nd dose of pembrolizumab by 3 weeks and a 4th patient will be accrued. If there are two patients in the initial cohort with non-hematologic toxicities grade 3, or if hematological toxicity in two patients is grade 4 or higher, the second cohort will delay initiation of pembrolizumab until post operative day 35 after LITT. Conversely, if there are no non-hematologic adverse events (AEs) of grade 3 or higher, the investigators will proceed to cohort IB using the same dose of pembrolizumab given 7 days prior to surgery, then every 3 weeks. Similarly, feasibility and safety will be addressed as above in deciding whether or not to proceed to the next cohort.

The Phase II component of the study will consist of additional patients receiving pembrolizumab at the earliest tolerated time post LITT:

* 14 days post-op
* -7 days pre-op;
* 35 days post-opto achieve a total of 23 evaluable patients at the earliest tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma or gliosarcoma prior to registration by pathology report;
* The tumor must be confined to the supratentorial compartment
* The Formaldehyde Fixed-Paraffin Embedded tumor tissue block must be available to be sent for retrospective central pathology review after registration).
* History/physical examination within 7 days prior to registration
* Karnofsky performance status ≥ 60 within 7 days prior to registration
* Adequate Organ Function Laboratory Values

  * Absolute neutrophil count (ANC) ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥9.0 g/gL or ≥5.6 mmol/L, without recent transfusion
  * Creatine ≤1.7 x upper limit of normal (ULN) or Measure or Calculated creatinine clearance ≥ 60.0mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)
  * Total bilirubin ≤ 1.5 x ULN or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN or ≤ 5 x ULN for subjects with liver metastases
  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Adequate hematologic function based on complete blood count (CBC)/differential within 7 days prior to registration defined as follows:

  * Absolute neutrophil count ≥ 1,500 cells/mm3;
  * Platelet count ≥ 100,000 cells/mm3
  * Hgb > 9 g/dL (can be achieved with transfusion)
* Adequate renal function within 7 days prior to registration defined as follows:

  * Blood Urea Nitrogen (BUN) ≤ 30 mg/dl and
  * Serum creatinine ≤ 1.7 mg/dl
* Adequate hepatic function within 7 days prior to registration defined as follows:

  * Total bilirubin (except patients with Gilbert's Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) ≤ 2.0 mg/dl and
  * Alanine Aminotransferase (ALT) and Aspartate Amino Transferase (AST) ≤ 2.5 x ULN
* The patient must have completed chemoradiation with Radiotherapy and Temozolomide of the primary tumor according to standards of care
* The treating physician expects that the patient will not require more than physiologic replacement dose of steroids defined as 4 mg of dexamethasone per day or its equivalent.
* Patients must have received no more than 3 prior therapies for Recurrent High Grade Glioma
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Tumor diameter in the plane perpendicular to LITT trajectory must be ≤ 6.0 cm in diameter
* It must be the surgeon's expectation that ≥ 90 of the tumor can be treated with LITT to the yellow thermal damage threshold (TdT) line (ie, 43 degrees for 2 min)
* Tumor must be Unifocal & Unilateral-Two enhancing nodules within the same FLAIR hyperintense region are still eligible; 1-2 secondary enhancing or non-enhancing lesions may be present as long as they have been radiologically stable for greater than or equal to 3 months.

Exclusion Criteria:

* Use of an immunotherapy such as a vaccine therapy, dendritic cell vaccine or intracavitary or convectional enhanced delivery of therapy in the past
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Severe, active co-morbidity defined as follows:

  * Unstable angina within the last 6 months prior to registration
  * Transmural myocardial infarction within the last 6 months prior to registration
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of ≥ 2 mm using the analysis of an EKG performed within 7 days prior to registration
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
  * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months prior to registration
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for tumor resection.
  * Known history of Tuberculosis
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive and worsen the patient's HIV symptoms.
  * Active connective tissue disorders, such as lupus or scleroderma, which in the opinion of the treating physician may put the patient at high risk for immunologic toxicity.
  * History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis
  * Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or Chronic Inflammatory Demyelinating Polyneuropathy, myasthenia gravis; systemic autoimmune disease such as Systemic Lupus Erythematosus, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease.
  * Of note, patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
  * Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
  * Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
  * Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
  * Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * Has known history of, or any evidence of active, non-infectious pneumonitis.
  * Has an active infection requiring systemic therapy?
  * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
  * Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
  * Has received prior therapy with an anti-Programmed Death 1 (PD-1), anti- Programmed Death-ligand 1 (PD-L1), or anti- Programmed Death-ligand 1 (PD-L2) agent.
  * Has a known history of Human Immunodeficiency Virus (HIV) (HIV ½ antibodies).
  * Has known active Hepatitis B (e.g., HbsAg reactive) or Hepatitis C (eg, HCV RNA [qualitative] is detected).
  * Has received a live attenuated vaccine within 30 days of planned start of study therapy.

    * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however Intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Patient must have < 1.0 cm midline shift pre-operative
* History of severe hypersensitivity reaction to any monoclonal antibody including pembrolizumab.
* Patients who cannot safely undergo MRI due to non-MRI compatible pacemaker, or other reason.
* Patients who have tumors for which the Gd-enhancing mass appears to be covered ≤ 90% using 2 catheters and assuming a 3.0 cm diameter based on pre-operative planning are unlikely to have adequate LITT and thus ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase I endpoint: Optimal timing of LITT with pembrolizumab | Up to 24 months after beginning Pembrolizumab
  Optimal timing of LITT with pembrolizumab
Phase II endpoint: Tumor Response | Up to 24 months after beginning Pembrolizumab
  Response rates for the Phase II component will be calculated and compared to historical controls using chi-square tests or Fishers exact tests.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 24 months after beginning Pembrolizumab
  PFS, defined as time from diagnosis to documented progression
Overall survival (OS) | Up to 24 months after beginning Pembrolizumab
  OS, defined as time from diagnosis to death
The proportion of patients who achieve progression free survival at 6 months (PFS6) | Up to 6 months after diagnosis
  PFS6, Proportion of patients who do not progress at 6 months
The proportion of patients who achieve progression free survival at 12 months (PFS12) | Up to 12 months after diagnosis
  PFS12, Proportion of patients who do not progress at 12 months
The proportion of patients who achieve progression free survival at 24 months (PFS24) | Up to 24 months after diagnosis
  PFS24, Proportion of patients who do not progress at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Hodges, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States